CLINICAL TRIAL: NCT02810886
Title: Prospective Evaluation of 68Ga-PSMA-ligand PET-CT for Recurrence Detection of Prostate Cancer and Its Impact on Patient Management
Brief Title: Prospective Evaluation of 68Ga-PSMA PET-CT for Recurrence Detection of Prostate Cancer and Its Impact on Patient Management
Acronym: ProsPERo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Recent publications demonstrating the clinical interest in performing 68Ga-PSMA for recurrence detection of prostate cancer patients with biochemical relapse
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-PROS-PROSPERO-2016
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancers
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single, arm exploratory (Experimental): Patients will undergo a 68Ga-PSMA PET/CT within 1 month after routine imaging diagnostic work-up.
  Interventions: Drug: 68Ga-(HBED-CC)-PSMA

INTERVENTIONS:
Drug: 68Ga-(HBED-CC)-PSMA — 68Ga-PSMA-ligand intravenous administration duration is around one minute. Once the patient is injected, the tracer needs 60 minutes to be evenly distributed through the body. PET/CT images will then be performed.
  Other Names: 68Ga-PSMA; 68Ga-DKFZ-PSMA-11; 68Ga-PSMA-ligand

SUMMARY:
Single arm, phase II exploratory trial to prospectively evaluate the impact of 68Ga-PSMA-PET/CT on the therapeutic management of patients with biological recurrent prostate cancer and negative, equivocal or oligometastatic disease after routine imaging diagnostic work-up.

DETAILED DESCRIPTION:
68Ga-PSMA-ligand PET-CT is a recently developed molecular imaging technique. It is based on the prostate specific membrane antigen (PSMA), a transmembrane protein with a large extracellular domain which is over-expressed on prostate cancer cells surface. Initial experiments used a ligand to the extracellular epitope of PSMA and labelled it with the isotope 68Ga, a positron emitter (68Ga-PSMA-HBED-CC) 5.

Recently published data based on more than 300 patients show recurrence detection rates and tumour to background ratios higher than choline PET-CT, even at low Prostate Specific Antigen (PSA) levels (sensitivity of 70% in PSA<2ng/ml) 6,7. False-positive PSMA findings are not yet reported.

The therapeutic management of biochemical recurrence in prostate cancer depends on the localisation and the extent of the recurrent disease.

In this study, the hypothesis is that 68Ga-PSMA-ligand PET-CT, through its high diagnostic accuracy has a significant impact on the therapeutic management of patients with biochemical recurrence.

Primary objective:

To prospectively evaluate the impact of PSMA-PET/CT on the therapeutic management of patients with biological recurrent prostate cancer and negative, equivocal or oligometastatic disease after routine imaging diagnostic work-up.

The treatment management decision will be recorded at the urologic tumor board (UTB) before and after the PSMA-PET/CT result. Rate of decision change will be calculated.

Secondary objective(s)

1. To compare detection rates of PSMA PET/CT and Routine Imaging Workup
2. To search for a predictor of a positive PET scan
3. To assess diagnostic value of PSMA-PET/CT
4. To assess PSA response after targeted treatment for oligometastatic disease.
5. To evaluate the delay to start of Androgen Deprivation Therapy (ADT) from the UTB decision.
6. To evaluate the time to PSA progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Histologically-proven prostate adenocarcinoma.
* Biochemical recurrence (BCR) after local treatment with radical curative intent based on PSA values 1:

  * Following Radical Prostatectomy +/- Radiotherapy: a serum PSA increase confirmed by a second PSA measurement higher than the first one with a value of 0.2 ng/mL or more within minimum of one week.
  * Following primary Radiotherapy: PSA value of 2 ng/ml above the nadir.
  * A continued rise in PSA level despite treatment with curative intent.
* Patients with negative, inconclusive or oligometastatic disease on the Routine Imaging Workup and susceptible to be treated with curative radical intent (salvage treatment).

  * Routing Imaging Workup exams are accepted when performed within 1 month before PSMA-PET/CT (this includes WB-MRI, prostatic/pelvic MRI, and/or Bone Scintigraphy).
* Patient treatment strategy based on routine diagnostic work-up needs to be recorded after discussion at the Urologic Tumor Board and available before the PSMA PET/CT.
* ECOG performance status ≤ 2
* Signed informed consent prior to any study related procedure.

Exclusion Criteria:

* Previous malignancy other than Prostate Cancer (except basocellular or squamous cell skin cancer).
* Patients treated with palliative chemotherapy or new hormonal therapies like Abiraterone/Enzalutamide.
* PSA rise while on active treatment (LHRH-agonist, LHRH-antagonist, anti-androgen, maximal androgen blockade, oestrogen). A minimal time window of 1 month is required.
* Medical castration with Testosterone < 50 ng/dl (1.7 nmol/L).
* Metastatic patients before inclusion not considered for targeted therapy.
* Previous treatment with isotopes (Radium, Samarium, Strontium, etc.)
* All medical conditions that might interfere with the correct performance of imaging scans.
* Known allergy/sensitivity to 68Ga or HBED-CC coupled substance, or any of the ingredient(s) or excipient(s) of the study medication(s)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Changes in treatment management are defined as: • Shift to a different therapeutic strategy • Modification of the initial therapeutic strategy • No changes | 2 months

SECONDARY OUTCOMES:
Number of positive scans | 2 months
  * PSMA only positive
  * Routine Imaging only positive
  * Positive in both
Correlation of positivity with: | 2 months
  * PSA value at the time of imaging
  * PSA doubling time
  * Gleason score
Reference diagnosis | 6 months
  * Histology when available.
  * Normalisation of PSA level after ablative therapy.
  * Morphological and/or biochemical evolution when no target treatment is given.
A confirmed PSA response is defined as ≥ 30% reduction of the blood level, compared to the baseline value, confirmed by a second PSA value 4 or more weeks later. PSA responses will be evaluated at for up to 6 months | 6 months
Androgen Deprivation Therapy (ADT) free survival: time from final Urologic Tumour Board treatment decision to start of ADT treatment during the follow up period of 6 months | 6 months
Time to prostate specific antigen (PSA) progression according to Prostate Cancer Clinical Trials Working Group criteria | 3 months
  * In case of decline from baseline: record time from final Urulogic Tumor Board treatment decision to first PSA increase that is ≥25% and ≥ 2 ng/ml above the nadir OR that is ≥25% above the pretreatment PSA value and which is confirmed by a second value 3 or more weeks later.
  * In case of no decline from baseline: PSA increase that is ≥25% and ≥ 2 ng/ml after 3 months if baseline PSA is ≥2 ng/ml. PSA increase that is ≥25% after 3 months if baseline PSA is < 2 ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Artigas, MD, Study Chair — Jules Bordet Institute

IPD SHARING:
Plan to Share IPD: No